CLINICAL TRIAL: NCT06885099
Title: Ease of Use Study of the FemPulse System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP013
Record Dates: First submitted 2025-02-11; First posted 2025-03-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Overactive Bladder (OAB)
Keywords: neuromodulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Subjects receiving the FemPulse System (Experimental): Subjects to receive the FemPulse System consisting of a non-implanted, vaginal electrical stimulation device (Ring) and other patient accessories.
  Interventions: Device: FemPulse System

INTERVENTIONS:
Device: FemPulse System — Subjects to receive the FemPulse System consisting of a non-implanted, vaginal electrical stimulation device (Ring) and other patient accessories.

SUMMARY:
The objective of the study is to demonstrate that the FemPulse System can be used as indicated

DETAILED DESCRIPTION:
The objective of the study is to demonstrate that the FemPulse System can be used as indicated in the Patient and Clinician Instructions for Use (IFU), as applicable.

ELIGIBILITY:
Key Inclusion Criteria:

1. Females, defined as a person with a cervix, ≥21 years old, with OAB symptoms, as confirmed by a physician. OAB is defined by urinary urgency, usually with urinary frequency and nocturia, with or without urgency urinary incontinence with symptoms .
2. Able to read, comprehend, and reliably provide informed consent and study-related information.
3. Willing and able to comply with study required procedures and visits

Exclusion Criteria:

1. Any significant pain, neurologic, psychological condition or other factors, that in the investigator's judgment, might confound the protocol study assessments, and adherence to the protocol.
2. Has a metal pelvic implant or an active implantable medical device, including but not limited to a cardiac pacemaker, cardioverter-defibrillator or neurostimulator 3 History of a cardiac condition including, but not limited to, clinically significant abnormal ECG or arrhythmia that may interfere with study participation as determined by investigator.

4. Systemic condition or disease that may interfere with study participation or not an appropriate study candidate, as determined by study investigator.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, defined as a person with a uterus and cervix.
Enrollment: 11 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Patient Usability of System | 2 days
  A survery will be conducted to determine the overall usability of the system

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — FemPulse Corporation
Locations (1):
- Holy Cross Women's Hospital, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No